CLINICAL TRIAL: NCT03384303
Title: Changes in Incretines, Gut Hormones and Bile Acids After Roux-en-Y Gastric
Brief Title: Changes in Incretines, Gut Hormones and Bile Acids After Roux-en-Y Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Principal Investigator, Frits Berends, Head of research department bariatric surgery, Rijnstate Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014-1359
Record Dates: First submitted 2017-12-04; First posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Morbid Obesity
Keywords: Incretines; Bile acids; Gut hormones; Limb lengths; Biliopancreatic limb; Bariatric surgery; Gastric bypass
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBPL-RYGB (Other)
  Interventions: Other: Standardized meal test
- S-RYGB (Other)
  Interventions: Other: Standardized meal test

INTERVENTIONS:
Other: Standardized meal test — Preoperatively and postoperatively standardized meal test

SUMMARY:
Obesity is an increasing world wide problem. Moreover, the increase in patients who are considered morbidly obese is even higher (Sturm et al, Healt Aff 2004). Conservative approaches such as diets or medication are unsuccessful in the majority of the patients. Additionally, (morbid) obesity leads often to cardiovascular diseases, such as hypertension, dyslipidemia and type 2 diabetes (T2DM). When patients need insulin to regulate their glucose levels, their weight is even more difficult to control. Therefore, bariatric procedures are increasingly performed, with over 8.000 procedures in the Netherlands in 2013. The two most performed types of bariatric surgery in the Netherlands are the Laparoscopic Roux-en-Y Gastric Bypass (LRYGB) and the Laparoscopic Sleeve Gastrectomy (LSG). Within the LRYGB there are different variants available. In a recently initiated randomized controlled trial (RCT) from our centre, a comparison between two variants of RYGB was performed. In this RCT our standard RYGB (s-RYGB:alimentary limb (AL) of 150cm; biliopancreatic limb (BPL) of 75cm) was compared with a RYGB with an long BPL (LBPLRYGB:AL of 75cm and a BPL of 150cm). A LBPLRYGB might improve weight loss and reduction after surgery. The exact mechanism of action is still not fully understood. Stomach volume is decreased and satiety levels often increase, probably due to changes in incretin levels. Passage of foods through the gastrointestinal tract are altered after RYGB. A possible explanation might be found in different levels of incretins (such as GLP-1, PYY and ghrelin) and bile acids (FGF-19 and FGF-21) after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* General guidelines for bariatric surgery according to Fried (Fried et al, Obes Surg 2007).
* Age > 18 years
* Patients must be able to adhere to the study visit schedule and protocol requirements
* Patients must be able to give informed consent and the consent must be obtained prior to any study procedures
* Patients who are planned for a LRYGB

Exclusion Criteria:

* Binge-eating or associated eating disorder
* Active drug or alcohol addiction
* Pregnancy and when giving breast feeding
* A medical history of bariatric surgery
* Patients with a language barrier which can inhibit patients to follow the correct medical advice
* Any kind of genetic disorder that can inhibit patients to follow the correct medical advice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline incretine levels during a standardized meal test four weeks after surgery. | Preoperatively and four weeks after surgery
Change from baseline gut hormone levels during a standardized meal test four weeks after surgery. | Preoperatively and four weeks after surgery
Change from baseline bile acid levels during a standardized meal test four weeks after surgery. | Preoperatively and four weeks after surgery

IPD SHARING:
Plan to Share IPD: No